CLINICAL TRIAL: NCT02750436
Title: A Prospective Randomized Comparison of Ultrasound Versus Fluoroscopic Guidance for Sacral Lateral Branch Blocks
Brief Title: A Comparison of Ultrasound Versus Fluoroscopic Guidance for Sacral Lateral Branch Blocks
Acronym: USGSLBB
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Montreal General Hospital (Other)
Responsible Party: Principal Investigator, Roderick Finlayson, Professor Department of Anesthesia, Montreal General Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 15-544MUHC
Record Dates: First submitted 2016-04-17; First posted 2016-04-25 (Estimated); Last update posted 2017-03-27 (Actual); Status verified 2017-03

CONDITIONS: Back Pain
MeSH Terms: conditions — Back Pain

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Ultrasound guided (Experimental): Ultrasound guided sacral lateral branch block
  Interventions: Device: Ultrasound guided
- Fluoroscopy guided (Active Comparator): Fluoroscopically guided sacral lateral branch block
  Interventions: Device: Fluoroscopy guided

INTERVENTIONS:
Device: Ultrasound guided — This group will be treated using an ultrasound imaging device
  Other Names: Ultrasound guided sacral lateral branch block
  Arms: Ultrasound guided
Device: Fluoroscopy guided — This group will be treated using a fluoroscopy imaging device
  Other Names: Fluoroscopically guided sacral lateral branch block
  Arms: Fluoroscopy guided

SUMMARY:
Sacral lateral branch blocks are used for the diagnosis and treatment of sacroiliac joint pain. This study will compare ultrasound and fluoroscopy guidance for sacral lateral branch blocks. Outcomes examined will include performance times and success rates.

ELIGIBILITY:
Inclusion Criteria:

* Any consenting patient over 18 years of age, undergoing a diagnostic sacral lateral branch block for suspected sacroiliac joint related pain.

Exclusion Criteria:

* Inability to consent, iodine or lidocaine allergy, pregnancy, coagulopathy (as defined by an international normalized ratio over 1.4, platelets under 100,000, or a documented bleeding disorder) and inability to visualize the target areas necessary for sensory testing (posterior superior iliac spine, dorsal aspect of SIJ) under ultrasound guidance.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2016-04-25 (Actual); Primary Completion 2016-07-30 (Actual); Study Completion 2016-07-30 (Actual)

PRIMARY OUTCOMES:
Performance time | Duration of procedure (less than 20 minutes)
  Block performance time will be measured from the time the first image is acquired, until the last injection is completed. Typical performance time are expected to be less than 20 minutes for both groups.

SECONDARY OUTCOMES:
Change in pain numerical rating score from baseline | Baseline and 20 minutes after procedure
  The extent of anesthesia provided by the blocks will be assessed by probing structures known to be innervated by the lateral branches and L5 posterior root. Two pain measurements will be undertaken, before and 20 minutes after the injections. Pain reports will be quantified by using a numerical rating score.

CONTACTS AND LOCATIONS:
Overall Officials: Roderick J Finlayson, MD, Principal Investigator — McGill University Health Centre/Research Institute of the McGill University Health Centre
Locations (1):
- Montreal General Hospital, Montreal, Quebec, Canada

IPD SHARING:
Plan to Share IPD: No